CLINICAL TRIAL: NCT04012554
Title: The Feasibility and Safety of Avoiding Chest Tube Placement After Video-assisted Thoracoscopic Surgery (VATS）of the Lung
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xueying Yang (Other)
Responsible Party: Sponsor-Investigator, Xueying Yang, professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-2019-HY-023
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Lung Diseases
Keywords: Postoperative pain; Avoiding chest drainage placement; Hospital cost
MeSH Terms: conditions — Lung Diseases; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial.The main study content is the feasibility and safety of avoiding chest tube placement after VATS of the lung,participants were divided into experimental group and control group.Avoiding chest tube placement after VATS of the lung in the experimental group.Indwelling thoracic drainage tube after VATS of the lung in the control group.
Who Masked: Outcomes Assessor
Masking Description: This is a randomized controlled trial.Partcipants,Care Provider, and Investigator all know the grouping situation.The Investigator collect the information and observation indicators of the two groups of participant and send the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- avoiding chest drainage tube placement after resection of lung (Experimental): This group of patients underwent avoiding chest drainage tube placement after VATS of the lung.
  Interventions: Procedure: avoid chest drainage tube placement after video-assisted thoracoscopic wedge resection of lung
- indewlling chest drainage tube after resection of lung (Other): This group of patients underwent indewlling chest drainage tube after VATS of the lung.
  Interventions: Procedure: Indewlling chest drainage tube after video-assisted thoracoscopic wedge resection of lung

INTERVENTIONS:
Procedure: avoid chest drainage tube placement after video-assisted thoracoscopic wedge resection of lung — Avoiding chest drainage tube placement after VATS of the lung in the experiment group.
  Arms: avoiding chest drainage tube placement after resection of lung
Procedure: Indewlling chest drainage tube after video-assisted thoracoscopic wedge resection of lung — Indewlling chest drainage tube after VATS of lung in the control group.
  Arms: indewlling chest drainage tube after resection of lung

SUMMARY:
This is a prospective randomized controlled trial.The main study content is the feasibility and safety of avoiding chest tube placement after Video-Assisted Thoracoscopic Surgery lung disease,participants were randomly divided into experimental group and control group.Avoiding chest tube placement after VATS of the lung in the experimental group.Indwelling thoracic drainage tube after VATS of the lung in the control group.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial.The main study content is the feasibility and safety of avoiding chest tube placement after VATS of the lung,divided into experiment group and control group.Communicating with surgeon and patients who met the inclusion criteria,decided whether to enter the experimental group or control group. Experimental group avoid chest tube placement after VATS of the lung and control group indwell thoracic drainage tube after VATS of the lung.By collecting personal information of two groups of patients and the corresponding observation indicators to analyze whether the treatment of avoiding chest tube placement after VATS of the lung is more beneficial than the conventional indwell thoracic drainage tube after VATS of the lung,and it's safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

- 1.Age ranges from 18 to 75 years old,do the examination of chest CT showed pulmonary disease,no invasion of peripheral blood vessels and viscera,no pleural effusion and pericardial effusion.

2.Electrocardiogram, pulmonary function,color doppler ultrasound of the heart,arteries and veins of both lower limbs are normal,no potential infection was confirmed before surgery, no serious organic disease of the heart and lung,and no obvious operation contrain.

Exclusion Criteria:

* 1.The lungs continue to leak air preoperation more than six days. 2.The appearment of the hemothorax,empyema and chylothorax preoperative. 3.The appearment of the preoperative chest X-ray pulmonary atelectasis and pulmonary infection.

  4.The lungs leak air appears in the surgery. 5.Patients with severe cardiovascular and cerebrovascular accident after operation were terminated.

  6.Impaired lung function (forced expiratory volume in 1 second [FEV1]<60% predicted).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
operation time | 1 day
  From the beginnning of ansesthesia to the end of anesthesia
hospitalization expenses | 15 days
  the total cost of hospitalzation
postoperative complication rate | a month
  incidence of postoperative complications such as pneumothorax and hydrohorax
duration of postoperation pain | 10 days
  postoperative pain duration
VAS pain scores | 3 days
  the VAS pain score was given to patients and the pain scores were recorded at 6h,12h,24h,48h,and 72h postoperatively.The minimum score is 0 and the maximum score is 10.The high values represent a worse outcome.
the time of early ambulation after operation | 1 day
  the time from the patient's postoperative pushback to the first bedtime
postoperative extubation time | 1 day
  postoperative extubation time

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Yang, M.D., Principal Investigator — The Fourth Affiliated Hospital of China Medical University
Locations (1):
- The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
hospital cost and complications of postoperation
Supporting Information: Study Protocol
Time Frame: data will become available in the next six month
Access Criteria: Feasibility and Safety of Postoperative Management Without Chest Tube Placement After VATS pneumoresection
URL: http://link-springer-com-cd.vtrus.net/content/pdf/10.1007%2Fs00595-010-4346-5.pdf

REFERENCES:
- [Result] Nakashima S, Watanabe A, Mishina T, Obama T, Mawatari T, Higami T. Feasibility and safety of postoperative management without chest tube placement after thoracoscopic wedge resection of the lung. Surg Today. 2011 Jun;41(6):774-9. doi: 10.1007/s00595-010-4346-5. Epub 2011 May 28. PMID 21626321
- [Result] Holbek BL, Hansen HJ, Kehlet H, Petersen RH. Thoracoscopic pulmonary wedge resection without post-operative chest drain: an observational study. Gen Thorac Cardiovasc Surg. 2016 Oct;64(10):612-7. doi: 10.1007/s11748-016-0692-6. Epub 2016 Aug 10. PMID 27510705
- [Result] Li P, Shen C, Wu Y, Lai Y, Zhou K, Che G. It is safe and feasible to omit the chest tube postoperatively for selected patients receiving thoracoscopic pulmonary resection: a meta-analysis. J Thorac Dis. 2018 May;10(5):2712-2721. doi: 10.21037/jtd.2018.04.75. PMID 29997933
- [Result] Filosso PL, Sandri A, Guerrera F, Roffinella M, Bora G, Solidoro P. Management of Chest Drains After Thoracic Resections. Thorac Surg Clin. 2017 Feb;27(1):7-11. doi: 10.1016/j.thorsurg.2016.08.002. PMID 27865329
- [Result] Russo L, Wiechmann RJ, Magovern JA, Szydlowski GW, Mack MJ, Naunheim KS, Landreneau RJ. Early chest tube removal after video-assisted thoracoscopic wedge resection of the lung. Ann Thorac Surg. 1998 Nov;66(5):1751-4. doi: 10.1016/s0003-4975(98)00946-1. PMID 9875783
- [Result] Lu TY, Chen JX, Chen PR, Lin YS, Chen CK, Kao PY, Huang TM, Fang HY. Evaluation of the necessity for chest drain placement following thoracoscopic wedge resection. Surg Today. 2017 May;47(5):606-610. doi: 10.1007/s00595-016-1414-5. Epub 2016 Sep 29. PMID 27688029
- [Result] Watanabe A, Watanabe T, Ohsawa H, Mawatari T, Ichimiya Y, Takahashi N, Sato H, Abe T. Avoiding chest tube placement after video-assisted thoracoscopic wedge resection of the lung. Eur J Cardiothorac Surg. 2004 May;25(5):872-6. doi: 10.1016/j.ejcts.2004.01.041. PMID 15082297
- [Result] Deng B, Qian K, Zhou JH, Tan QY, Wang RW. Optimization of Chest Tube Management to Expedite Rehabilitation of Lung Cancer Patients After Video-Assisted Thoracic Surgery: A Meta-Analysis and Systematic Review. World J Surg. 2017 Aug;41(8):2039-2045. doi: 10.1007/s00268-017-3975-x. PMID 28289835
- [Result] Chiappetta M, Lococo F, Nachira D, Ciavarella LP, Congedo MT, Porziella V, Meacci E, Margaritora S. Digital Devices Improve Chest Tube Management: Results from a Prospective Randomized Trial. Thorac Cardiovasc Surg. 2018 Oct;66(7):595-602. doi: 10.1055/s-0037-1607443. Epub 2017 Oct 27. PMID 29078230